CLINICAL TRIAL: NCT04166422
Title: Virtual Reality and Video Games in Cardiac Rehabilitation Programs. A Randomized Controlled Trial
Brief Title: Virtual Reality and Video Games in Cardiac Rehabilitation Programs
Acronym: VirtualCORE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, Full Professor, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VIRTUAL CORE URJC
Record Dates: First submitted 2019-11-11; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Adherence, Patient; Physical Disability; Cardiovascular Diseases; Treatment Adherence; Satisfaction
MeSH Terms: conditions — Patient Compliance; Cardiovascular Diseases; Treatment Adherence and Compliance; Personal Satisfaction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional group (Active Comparator): Conventional rehabilitation treatment
  Interventions: Other: Cardiac rehabilitation program
- Experimental group (Experimental): Virtual reality plus conventional rehabilitation treatment
  Interventions: Other: Experimental intervention

INTERVENTIONS:
Other: Cardiac rehabilitation program — Aerobic treatment plus strength exercises
  Arms: Conventional group
Other: Experimental intervention — Aerobic treatment plus strengh exercises plus virtual reality
  Arms: Experimental group

SUMMARY:
Cardiovascular diseases (CVD) are the leading cause of morbidity and mortality in developed countries. The consequent healthcare costs in Europe alone are estimated at 196,000 million euros annually, approximately 54% of the total investment in health, resulting in productivity losses of 24% [1-3]. In recent years, the impact of CVD in non-Western countries has been growing [4,5]; therefore, prevention is presented as a primordial tool to improve quality of life and patient survival [6,7]. Cardiac rehabilitation (CR) is defined as a multidisciplinary program of clinical application of preventive measures for risk reduction and global and long-term care of the cardiac patient. In secondary prevention, it is shown to reduce the morbimortality by almost 50% in patients with heart disease. However, the participation of patients in cardiac rehabilitation remains low, especially among the following groups: the elderly, women and patients with a low socioeconomic profile. According to the latest Euroaspire V data, participation in CR programs in Spain is around 50%. The Reureca registry reports that only 10% of patients with a CR indication attend the programs. Therefore, new technologies within the health field, specifically within cardiac rehabilitation programs through the use of virtual reality (VR) and video games, are shown as promising aids with the aim of increasing adherence, satisfaction with programs and participation rates, offering the ability to perform physical exercise [8-11]. Virtual reality is a simulation of a real or imaginary environment created by a computer system, which allows the user to feel immersed and to interact with objects in that environment [12-14]. Thus, the basic elements that constitute a VR system are simulation, interaction and immersion [15]. Moreover, the creation of more adaptable and accessible videogame platforms has meant that the phenomenon of technological expansion can be understood not only as a form of leisure but also as an important means of learning and skills training, especially in people with motor, cognitive and sensory (neurological and non-neurological) deficits [16]. In contrast to traditional CR procedures, which can be repetitive, causing a loss of interest on the part of patients, video games and VR systems offer the opportunity to participate in enjoyable tasks with a therapeutic purpose through physical interaction with the game. The design of exercise-based videogames (exergames) provides the possibility of practicing physical skills in an entertaining way and of adjusting the game according to the abilities of the subject and the level of intensity. In addition, it is known that the level of enjoyment of an activity has been identified as one of the predictive factors of the effectiveness of an exercise program, and for this reason, interactive technology based on exercise is becoming the all-time most popular strategy for the implementation of physical activity [17-23]. It is important to emphasize that VR allows the creation of environments suitable for activities related to CR. The users of these systems can develop simulated tasks and activities in a safe way, since the clinicians have the capacity to control the duration and intensity of the exercise and, in this way, to control and supervise the delivery of stimuli in the virtual environment [24]. Furthermore, knowledge of results regarding the performance of the task in real time, gained through extrinsic feedback, as well as the playful nature of the activities proposed through VR and videogame devices, generates a competitiveness and challenge component that further increases the degree of patient motivation. In this regard, Klasen et al. [25] point out that this increase in motivation is related to the influence of videogames on activation of the mesolimbic dopaminergic pathways and their repercussions on the reward system of the brain. All this promotes active participation on the part of the patient and thus increases adherence to the rehabilitation treatment. The aim of the present work is to carry out a RCT to provide information on the application of VR and videogame systems within CR programs in patients with cardiac diseases.

ELIGIBILITY:
Inclusion Criteria:

* either male or female;
* agegreater than 18 years;
* a diagnosis of CVD confirmed by a Cardiologist;
* information available on risk stratification, Killip level and functional class (NYHA), level according to the Canadian Cardiovascular Society Scale or the Goldman Physical Activity Scale;
* information available on METS in ergometry and ejection fraction and compliance with the indications described in relation to CR.

Exclusion Criteria:

* pregnancy or planned pregnancy,
* high cardiovascular risk,
* the presence of a pacemaker,
* conditions that make it difficult or impossible to use VR, such as the presence of visual or auditory deficiencies, learning problems, cognitive deterioration, psychiatric pathology or the use of support products for walking or standing,
* the presence of other serious neurological, musculoskeletal or lung diseases,
* uncompensated metabolic disorders,
* previous cardiorespiratory arrest
* a history of photosensitive epilepsy due to the use of video games.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-11-11 (Estimated); Study Completion 2021-11-11 (Estimated)

PRIMARY OUTCOMES:
METS in ergometry and ejection fraction | 8 weeks
  Ergometry is a science that measures work. A device that can be used to measure work is called an ergometer

SECONDARY OUTCOMES:
6 minute walking test | 8 weeks
  How long, in meters, walk a patients in 6 minutes
Functional Independence Measure (MIF) | 8 weeks
  This is an instrument that evaluates the inability of patients with functional restrictions of various causes; it quantitatively evaluates the care demand of a person for performing motor and cognitive tasks of daily living.
Short Form Quality of Life (SF36) | 8 weeks
  The Short Form (36) Health Survey is a 36-item, patient-reported survey of patient health.

OTHER OUTCOMES:
Adherence to the therapy sessions | 8 weeks
  the attendance rate (%) for therapy sessions
Satisfaction questionaire | 8 weeks
  which evaluate the level of satisfaction regarding the care and quality of the service received and the level of fulfillment of the patient's expectations regarding the treatment administered

CONTACTS AND LOCATIONS:
Locations (1):
- Roberto Cano de la Cuerda, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No